CLINICAL TRIAL: NCT00427141
Title: A Three-part First Time in Human Study to Evaluate Safety, Tolerability, Pharmacokinetics and Food Effect of Single Oral Doses of GSK580416 in Healthy Adult Subjects
Brief Title: A Three-Part Study Of GSK580416 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OPS106400
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Respiratory Tract Infection; Infections, Bacterial
Keywords: tolerability,; pharmacokinetics,; first time in human,; food effect; safety,
MeSH Terms: conditions — Respiratory Tract Infections; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK580416

SUMMARY:
Studies for GSK580416 have been completed in rats and dogs. The main toxic effects seen in animals affected the digestive system and blood cells. Study OPS106400 will be the first administration of GSK580416 in humans. Parts A and B of this study will examine the safety, tolerability, and pharmacokinetics of increasing single doses of GSK580416 with reference to placebo. Part C of the study will assess the effect of food on the safety, tolerability, and pharmacokinetics of a single dose of GSK580416 in healthy subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy as determined by a physician
* Healthy male or female of non-child bearing potential between 18 and 55 years of age (inclusive)
* Body weight > = 50 kg and BMI between 19 and 30 kg/m2 (inclusive)

Exclusion criteria:

* Positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody with 3 months of screening
* Male and female subjects not willing to follow study specified contraceptive methods
* Subjects taking any recreational drugs
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* Has participated in a clinical trial and have not received a drug within 30 days before the dose of study drug
* Has exposed to more than 4 new chemical entities within 12 months before the first dosing day
* Use of prescription or over-the-counter medications within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
* Use of St. John's Wort within 28 days before the first dose of study drug
* Subjects not willing to follow study specified life style restrictions
* Blood donation in excess of 500 mL within a 56 days period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Safety assessments (adverse event, ECG and vital sign) will be performed during the study. Blood samples to determine drug levels in the body will be collected during the study. | during the study

SECONDARY OUTCOMES:
Blood samples to determine drug levels in the body will be collected during the study. | during the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia